CLINICAL TRIAL: NCT01839149
Title: A Phase 2, Enriched-enrollment, Randomized-withdrawal, Double-blinded, Placebo-Controlled Study to Assess the Efficacy, Tolerability, and Safety of Intranasal Oxytocin in Subjects With Chronic Migraine
Brief Title: TI-001 (Intranasal Oxytocin) for Treatment of High Frequency Episodic Migraine and Chronic Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trigemina, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRIG-05
Record Dates: First submitted 2013-04-17; First posted 2013-04-24 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: High Frequency Episodic Migraine and Chronic Migraine
Keywords: Refractory Chronic Migraine; Medically Intractable Chronic Migraine; Oxytocin; Intranasal oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TI-001 (intranasal oxytocin) (Experimental): TI-001 is intranasal oxytocin
  Interventions: Drug: TI-001
- Placebo (Placebo Comparator): Placebo for TI-001 is the same intranasal formulation without oxytocin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TI-001 — TI-001 is intranasal oxytocin
  Other Names: Intranasal oxytocin
  Arms: TI-001 (intranasal oxytocin)
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the use of oxytocin, given as a nasal spray, for treatment of high frequency episodic migraine and chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 to 65 years with primary diagnosis of high frequency episodic migraine or chronic migraine.

Exclusion Criteria:

1. Known allergy to oxytocin
2. History of addictive behavior (eg, alcoholism, drug abuse) or severe mood disorder
3. History of clinically significant, functionally impairing cardiovascular or pulmonary disease or any other disease that might confound study results
4. Have basilar or hemiplegic migraines
5. Have substantial cognitive or memory impairment due to any cause (eg, Alzheimer's or dementia)
6. Have a nasal obstruction due to any cause
7. Are pregnant or breast feeding
8. Require ongoing use of steroidal or nonsteroidal anti-inflammatory drugs
9. Are unable or unwilling to provide informed consent or to follow study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-05; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mean change of migraine days | Baseline and 28 days of treatment
  Baseline is the 28-day screening period before study drug administration

SECONDARY OUTCOMES:
Mean change of moderate or severe headache days | Baseline and 28 days of treatment
Proportion of subjects experiencing a ≥50% reduction in migraine days | Baseline and 28 days of treatment
Mean change in days using rescue medication | Baseline and 28 days of treatment
Proportion of subjects experiencing a reduction in headache severity and pain score 2 hours after dosing | Baseline and 28 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Izumi, PhD, Study Director — Trigemina, Inc
Locations (6):
- Australia (3):
  - Fitzroy
  - Prahran
  - Sherwood
- Santiago, Chile
- New Zealand (2):
  - Tauranga
  - Wellington